CLINICAL TRIAL: NCT02079025
Title: Multi-Center Trial of High-resolution Transrectal Ultrasound Versus Standard Low-resolution Transrectal Ultrasound for the Identification of Clinically Significant Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exact Imaging (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-UHR-002
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Prostatic Neoplasms; Prostate Cancer; Cancer of the Prostate
Keywords: Prostate Biopsy; Ultrasound guided biopsy of the prostate; High-resolution ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LR-TRUS (Active Comparator): Low-resolution transrectal ultrasound guided prostate biopsy (standard of care)
  Interventions: Device: Standard ultrasound guided prostate biopsy
- UHR-TRUS (Experimental): Ultra-high resolution transrectal ultrasound guided prostate biopsy
  Interventions: Device: High-resolution ultrasound guided prostate biopsy

INTERVENTIONS:
Device: High-resolution ultrasound guided prostate biopsy — Ultrasound guided prostate biopsy using ultra-high resolution ultrasound system
  Other Names: ImagistxProstate Urology Ultrasound System
  Arms: UHR-TRUS
Device: Standard ultrasound guided prostate biopsy — Ultrasound guided prostate biopsy using standard of care ultrasound system
  Arms: LR-TRUS

SUMMARY:
This trial uses a ultra high-resolution ultrasound system and specialized transducer, intended for use in prostate imaging. The system's image resolution is significantly better than the standard of care, due to its higher frequency. This allows the system to visualize suspicious areas and structures, and for greater accuracy for guided biopsy.

The primary objective of this study is to demonstrate that ultra high-resolution transrectal ultrasound (UHR-TRUS) is superior to conventional low-resolution transrectal ultrasound (LR-TRUS) in detecting clinically significant cancer among men without known prostate cancer and with an indication for prostate biopsy.

The secondary objective of this study is to compare the difference in the rate of detection of clinically significant cancer between LR-TRUS and UHR-TRUS, from before investigator training to after investigator training.

The tertiary objective for the investigation is to compare the combined sensitivity and specificity in determining cancer detection overall for image-guided biopsy in UHR-TRUS vs. LR-TRUS.

DETAILED DESCRIPTION:
This is a two-arm multi-centre randomized trial of LR-TRUS versus UHR-TRUS for guided prostate biopsies in men with no known history of prostate cancer. This trial will enroll a minimum of 800 and a maximum of 2000 patients with regular interim analyses to determine the trial's final sample size. These numbers are based on predictive probabilities of trial success.

The investigation is designed as a comparative non-blinded analysis of LR-TRUS vs. UHR-TRUS. Participants will be randomized to either high-resolution or low resolution ultrasound with an equal chance of being in either group. The randomization scheme will be stratified by centre.

When a subject arrives at the institution for his biopsy, the Study Coordinator opens a sealed envelope that indicates to the study participant and physician whether the procedure will be performed using LR-TRUS or UHR-TRUS.

All subjects have an indication for prostate biopsy, and thus, inclusion of a non-treatment group would necessitate a group of men not to receive standard of care. As such, there is no control group in the subject population.

Procedures in the study are:

* obtaining informed consent for the subject
* collecting pre-biopsy information and recording it on the case report form (CRF)
* perform biopsy procedure
* record biopsy details in CRF
* prepare biopsy specimens for pathology

Data from CRFs will be stored in a proprietary database that is accessed by a web-based interface, where access is limited to those with login and password. No subject-identifiable information will be entered in the database.

The primary endpoint is the detection of clinically significant prostate cancer, i.e., the number of men with clinically significant prostate cancer determined by pathology review among all men randomized and biopsied. Pathological analysis on 12-core biopsy samples will be the only mechanism used to determine if study subjects have prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* All men > 40 years age and <80 years of age with an indication for a prostate biopsy will be offered inclusion in the study. Typical indications for biopsy include abnormal PSA (prostate specific antigen) and/or abnormal DRE (digital rectal exam).
* PSA<50
* Clinical stage < cT3

Exclusion Criteria:

* Men with a history of prostate cancer
* Men undergoing TRUS-guided prostate biopsy in the OR under anesthesia
* Men with known prostate volume (from prior imaging) of > 60cc
* Men with anorectal abnormalities preventing TRUS-guided prostate biopsy
* Men who are unable to provide their own informed consent

Ages: 40 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1676 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Johns Hopkins Brady Urological Institution, Baltimore, Maryland
  - Urology of Virgina, Virginia Beach, Virginia
- Canada (3):
  - Prostate Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre de Recherche sur le Cancer ("CRCEO"), Québec, Quebec

REFERENCES:
- [Derived] Rohrbach D, Wodlinger B, Wen J, Mamou J, Feleppa E. High-Frequency Quantitative Ultrasound for Imaging Prostate Cancer Using a Novel Micro-Ultrasound Scanner. Ultrasound Med Biol. 2018 Jul;44(7):1341-1354. doi: 10.1016/j.ultrasmedbio.2018.02.014. Epub 2018 Apr 4. PMID 29627083

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LR-TRUS | UHR-TRUS
Started | 839 | 837
Completed | 839 | 837
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LR-TRUS | UHR-TRUS | Total
Number analyzed (Participants) | 839 | 837 | 1676
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.67) | 62.7 (8.66) | 62.7 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 839 | 837 | 1676
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 279 | 272 | 551
  United States | 560 | 565 | 1125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant Prostate Cancer
Description: Pathology analysis of prostate biopsy is reviewed for indication of clinically significant prostate cancer. Interim analyses are planned beginning when 800 patients have been enrolled and after every additional 200 patients are enrolled up to the maximum sample size of 2000 patients.
Time Frame: First visit (a patient's involvement in the trial is complete following his biopsy).
Population: Intent To Treat includes all subjects, Per Protocol includes only subjects without protocol deviations.
Measure: Number; unit: percentage of participants with csPCa
Arm/Group | LR-TRUS | UHR-TRUS
Number analyzed (Participants) | 839 | 837
percentage of participants with csPCa
  Intent to Treat | 36.6 | 34.6
  Per Protocol: number analyzed (Participants) | 823 | 286
  Per Protocol | 36.6 | 43.7

2. Secondary Outcome: Improvement of an Investigator's Ability to Detect Clinically Significant Cancer Using UHR-TRUS Post-training When Compared to Pre-training
Description: Comparison of pre- and post-training percentage of participants found to harbor clinically significant prostate cancer within the UHR-TRUS arm of the trial
Time Frame: Pre-training refers to all biopsy procedures occurring between initial training and mid-trial PRI-MUS training. Post-training refers to all biopsy procedures performed after mid-trial PRI-MUS training.
Population: Pre and post-training detection rate for csPCa for the UHR-TRUS arm only (as investigators received additional training on this imaging modality)
Measure: Number; unit: Percentage of subjects with csPCa
Arm/Group | UHR-TRUS
Number analyzed (Participants) | 837
Percentage of subjects with csPCa
  Pre-Training: number analyzed (Participants) | 555
  Pre-Training | 32.4
  Post-Training: number analyzed (Participants) | 282
  Post-Training | 39.0

3. Secondary Outcome: Combined Sensitivity and Specificity in Determining Cancer Detection Overall for Image-guided Biopsy
Description: Pathology analysis of prostate biopsy is reviewed. Sensitivity of targeted biopsy for each arm will be calculated as the number of targeted biopsy that also found cancer among all targeted biopsies. Specificity of targeted biopsy for each arm will be calculated as the number of non-targeted biopsies that find no cancer among all non-targeted biopsies. Interim analyses are planned beginning when 800 patients have been enrolled and after every additional 200 patients are enrolled up to the maximum sample size of 2000 patients.
Time Frame: First visit (a patient's involvement in the trial is complete following his biopsy).
Measure: Number; unit: percentage of post-training samples
Units Other Than Participants: Post-training biopsy samples
Arm/Group | LR-TRUS | UHR-TRUS
Number analyzed (Participants) | 839 | 837
Number analyzed (Post-training biopsy samples) | 3372 | 3384
percentage of post-training samples
  Sensitivity | 38.0 | 60.8
  Specificity | 89.5 | 63.2

ADVERSE EVENTS:
Arm/Group | LR-TRUS | UHR-TRUS
Serious Adverse Events (participants affected / at risk) | 3/839 | 3/837
Other Adverse Events (participants affected / at risk) | 0/839 | 0/837
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LR-TRUS (N=839) | UHR-TRUS (N=837)
post-biopsy bacteremia (Infections and infestations) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No